CLINICAL TRIAL: NCT02696421
Title: Ramadan and Energy (RAMEE) Study
Brief Title: Ramadan and Energy Expenditure Study
Acronym: RAMEE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IREC 022
Record Dates: First submitted 2015-06-15; First posted 2016-03-02 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Energy Expenditure During Ramadan Fasting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Non diabetic, non obese
- Non diabetic obese
- Diabetic

SUMMARY:
Ramadan fasting entails abstinence from eating and drinking between dawn and sunset. During this month major changes in meal times and patterns, sleeping times and activity occur. Starvation is known to lead to a compensatory reduction in energy expenditure. However, the Ramadan fast is not synonymous with starvation as it involves intermittent periods of fasting followed by gorging. People who fast during Ramadan feel less energetic. However, little is known about the effects of this religious practice on energy metabolism. .

The aim of this study is to assess energy dynamics before and/or after and during Ramadan fasting in non-obese participants. Resting metabolic rate (RMR), thermic effect of food (TEF), active energy expenditure (AEE) and total energy expenditure (TEE) in free-living conditions will be measured . Indirect calorimetry will be used to assess RMR and TEF, doubly labeled water will be used to measure TEE and activity monitors will measure physical activity. In addition, body composition analysis will be performed by bio-electrical impedance. Blood sample will be taken to exclude medical factors affecting energy metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate.
* Age (18-70) years.
* BMI (20-30 kg/m2).
* Physically and mentally healthy.
* Consent form signed.

Exclusion Criteria:

* Any patients with significant health problem.
* Pregnant and lactating females.
* Smokers.
* Consumption of caffeine before tests.
* Patients who have had vigorous exercise for the last 12 hours before visit.
* Patients with diabetes treated with drugs known to alter the metabolic rate.
* Patients who had bariatric surgery.
* Patients with eating disorders.
* Patients with conditions known to affect energy expenditure
* Patients on medication know to alter EE (Thyroxine, anti-thyroid drugs, certain cold remedies)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 50 healthy non-obese (BMI: 20-30) subjects (age: 18-70) will be recruited. We will aim for equal representation of men and women.
  Physically and mentally healthy. Consent form signed.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Resting metabolic rate | 3 months
24 hour energy expenditure | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Derived] Lessan N, Saadane I, Alkaf B, Hambly C, Buckley AJ, Finer N, Speakman JR, Barakat MT. The effects of Ramadan fasting on activity and energy expenditure. Am J Clin Nutr. 2018 Jan 1;107(1):54-61. doi: 10.1093/ajcn/nqx016. PMID 29381798